CLINICAL TRIAL: NCT06923514
Title: Using Machine Learning to Analyze the Prediction and Correlation of Health Literacy, Stress and Quality of Life in Heart Failure Patients
Brief Title: Health Literacy, Stress and Quality of Life in Heart Failure Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: (1133)113A-63
Record Dates: First submitted 2025-03-18; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: Machine learning, health literacy, stress, quality of life.
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure is showing a trend of affecting younger individuals. Middle-aged heart failure patients are often the economic backbone of their families. Studies have also pointed out that approximately 38.5% of patients with acute heart failure are re-hospitalized within a year of discharge due to worsening symptoms. Patients with lower health literacy tend to have poorer health outcomes and higher re-hospitalization rates. However, there is limited research on the life and work stress, health literacy, and quality of life of middle-aged heart failure patients. Therefore, this study aims to use machine learning to analyze and predict the correlations between health literacy, stress, and quality of life in heart failure patients.

This research is a cross-sectional correlational study, adopting convenience sampling. The study subjects are cardiology patients aged 18-65 diagnosed with heart failure classified as NYHA II or above by specialists at a regional teaching hospital in northern Taiwan. Data collection took place in the outpatient and inpatient departments of cardiology and cardiothoracic surgery. Structured questionnaires were used for one-on-one interviews, including basic demographic information of heart failure patients, the Chinese version of the European Health Literacy Survey Questionnaire (HLS-EU-Q47), the Chinese version of the Brief Resilience Scale (BRS), the Perceived Stress Scale (PSS), and the Minnesota Living with Heart Failure Questionnaire (MLHFQ). Data will be recorded using Excel, and statistical analysis will be conducted using SPSS version 22. Descriptive statistics such as percentages, means, and standard deviations will be used to describe the demographic and variable distributions. Independent t-tests, ANOVA, and Pearson correlation coefficient will be used to analyze correlations between variables. Machine learning will be employed to analyze and predict quality of life factors in heart failure patients. It is hoped that the results of this study can provide references for nursing practice, help with clinical patient assessment, and improve the quality of care for patients.

ELIGIBILITY:
Inclusion Criteria:

* The study subjects are cardiology patients aged 18-65 diagnosed with heart failure classified as NYHA II or above by specialists at a regional teaching hospital in northern Taiwan

Exclusion Criteria:

* 1.severe mental disease.2. terminal stage of other disease such as cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2025-11-03 (Estimated)

PRIMARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire | one year
  Use the Chinese version of the Minnesota Heart Failure Quality of Life to assess quality of life.
  Use the Chinese version of the Minnesota Heart Failure Quality of Life Questionnaire.There are 21 questions in total, scored from 0 to 5, with a total score of 105. The higher the score, the more serious the impact of the disease on life.

SECONDARY OUTCOMES:
health literacy | one year
  Use the Chinese version of European Health Literacy Survey Questionnaire (HLS-EU-Q) to assess health literacy .
  Use the Chinese version of HLS-EU-Q.There are 47 questions in total. Based on a four-point Likert scale, Total score 0-50. 0-25 means Inadequate,26-33 means Problematic,34-42 means Sufficient,43-50 means Excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Hei-Fen Hwang, PhD, Study Director — Natinal Taipei University of Nursing and Health Sciencs
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuhn TA, Gathright EC, Dolansky MA, Gunstad J, Josephson R, Hughes JW. Health Literacy, Cognitive Function, and Mortality in Patients With Heart Failure. J Cardiovasc Nurs. 2022 Jan-Feb 01;37(1):50-55. doi: 10.1097/JCN.0000000000000855. PMID 34581712
- [Result] Jiang S, Zhang X, Li X, Li Y, Yang W, Yao Y, Fu L, Zhao M, Zang X. Exploring Health Literacy Categories in Patients With Heart Failure: A Latent Class Analysis. J Cardiovasc Nurs. 2023 Jan-Feb 01;38(1):13-22. doi: 10.1097/JCN.0000000000000889. Epub 2022 Jan 13. PMID 36508237
- [Result] Heo S, Kang J, Shin MS, Lim YH, Kim SH, Kim S, An M, Kim J. Physical Symptoms, Depressive Symptoms, and Quality of Life in Patients With Heart Failure: Cluster Analysis. J Cardiovasc Nurs. 2024 Jan-Feb 01;39(1):31-37. doi: 10.1097/JCN.0000000000001043. Epub 2023 Sep 29. PMID 37787730
- [Result] Gowani AAA, Low G, Norris C, Hoben M. Internal structure validity and internal consistency reliability of the Minnesota Living with Heart Failure Questionnaire: a systematic review protocol. BMJ Open. 2023 Nov 8;13(11):e076780. doi: 10.1136/bmjopen-2023-076780. PMID 37940148
- [Result] Cajita MI, Cajita TR, Han HR. Health Literacy and Heart Failure: A Systematic Review. J Cardiovasc Nurs. 2016 Mar-Apr;31(2):121-30. doi: 10.1097/JCN.0000000000000229. PMID 25569150